CLINICAL TRIAL: NCT03836443
Title: Lipid Metabolism, Lipotoxicity and Nonalcoholic Fatty Liver Disease: Implication of Postprandial Cytotoxic Lipids
Brief Title: Postprandial Lipotoxicity and Nonalcoholic Fatty Liver Disease
Acronym: LITONAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: D20180507
Record Dates: First submitted 2019-01-17; First posted 2019-02-11 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2023-04

CONDITIONS: Nonalcoholic Fatty Liver Disease (NAFLD)
Keywords: NAFLD, toxic lipids, postprandial lipotoxicity
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: A "western diet" meal (high saturated fat, high refined sugar, high fructose) will be administered in each group (800 kcal/meal) after an overnight fast.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NAFL patients (group 1) (Active Comparator): A "western diet" meal (high saturated fat, high refined sugar, high fructose) will be administered in each group (800 kcal/meal).
  Interventions: Other: western diet" meal
- NASH patients (group 2) (Active Comparator): A "western diet" meal (high saturated fat, high refined sugar, high fructose) will be administered in each group (800 kcal/meal).
  Interventions: Other: western diet" meal

INTERVENTIONS:
Other: western diet" meal — A "western diet" meal (high saturated fat, high refined sugar, high fructose) will be administered in each group (800 kcal/meal) after an overnight fast.

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD) is mainly considered a nutrition-related disease and life-style/diet interventions showed some promising results. But in spite of this, there are no available markers to efficiently guide interventions. the hypothesize put farth by the investigators is that NAFLD patients develop postprandial abnormalities of plasma lipids upon "western diet" challenge, more severe in steatohepatitis (NASH) than in pure steatosis (NAFL), promoting liver injury. Our study aims to evaluate the presence of toxic lipids (such as free-fatty acids, ceramides, diacylglycerols, sphingolipids) in postprandial state after ingestion of a "western diet" in NAFLD patients. Consecutive patients (group 1: NAFL patients; group 2: NASH patients) with biopsy-proven NAFLD (liver biopsy < 6 months) will be recruited during a period of 12 month. Blood samples will be drawn at fasting, 2hours, 4hours, 6hours and 8hours after ingestion of a "western diet" meal. Plasma lipid profiles using lipidomics, circulating markers of liver injury and inflammation will be analyzed. the investigators will also assess the hepatotoxicity of plasma from NAFL or NASH patients in-vitro.

DETAILED DESCRIPTION:
Factors driving progression from steatosis (NAFL) to steatohepatitis (NASH) in patients with non-alcoholic fatty liver disease (NAFLD) remain largely unknown. Considerable data now indicate that steatosis per se is not a hepatotoxic event and may represent in fact a protective mechanism against free fatty acid (FFA)-induced toxicity. the investigators previously showed that Kupffer cells from NASH mice accumulate more toxic lipids (ceramides, diacylglycerols, sphingolipids) enhancing their proinflammatory polarization. Therefore, "quality" of accumulating lipids rather than "quantity" may play a central role in NAFLD progression. This is a pilot comparative study aiming to evaluate the presence of toxic lipids (such as free-fatty acids, ceramides, diacylglycerols, sphingolipids) in postprandial state after ingestion of a "western diet" in NAFL and NASH patients. The secondary outcomes were: to evaluate the relationship between postprandial circulating lipids and markers of liver injury and proinflammatory cytokines; to evaluate hepatotoxicity of postprandial lipids in vitro. A total of 24 consecutive patients (group 1: 12 NAFL patients; group 2: 12 NASH patients) with biopsy-proven NAFLD (liver biopsy < 6 months) will be recruited. A dietary evaluation covering the 2 previous weeks will be performed. Detailed anthropometric data will be collected (body mass index, waist and hip circumferences, abdominal height, cutaneous skinfolds) and serum metabolic parameters (standard lipid profile, lipoprotein levels, fasting plasma glucose, insulin levels, C-peptide levels, hemoglobin A1c) will be evaluated. After a 12hours overnight fast, patients will undergo an oral "western diet" test consisting in the ingestion of a high saturated fat, high refined sugar, high fructose-meal called "western diet" (800 kcal/meal). Blood samples will be drawn at fasting and then 2, 4, 6 and 8hours after ingestion of the standard meal. Each time plasma and serum samples will be stored at -80°C for subsequent analysis. Lipidomics will be used to quantify each plasma lipid class (neutral lipids, phospholipids and fatty acid methyl esters). Serum levels of cytokines will be assessed using multiple assay technology. Markers of liver injury will be assessed (aminotransferases, Keratin 18 fragments, microRNA-122) in the serum. Hepatocytes will be cultured with plasma from NAFL or NASH patients, and incubated overnight. In vitro hepatotoxicity will be evaluated using TUNEL assay, MTT assay and LDH release assay. the investigators anticipate that inflammation together with hepatocyte death will occur in NAFLD patients who develop specific postprandial plasma lipid changes with an increase in toxic lipid levels. Such patients may develop more severe liver lesions (inflammation, fibrosis/cirrhosis) and benefit of interventions. Identification of a toxic plasma lipid profile may help choosing the adequate diet in order to prevent deleterious lipid formation. Identification of a toxic postprandial plasma lipid signature specific to hepatotoxicity may also serve to develop a discrimination index to be further validated in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

- histological proven NAFLD (liver biopsy <6 months); hospitalised or outpatients followed up for NAFLD; patients giving their consent for the study; patients covered by health insurance.

Exclusion Criteria:

* history of excessive alcohol consumption (>20 g/day for males and >10 g/day for females) or other cause of liver injury (viral hepatitis, autoimmune hepatitis, Wilson's disease, hemochromatosis, drug-induced hepatitis, or others); cirrhosis; ongoing hypolipemiant treatment; diabetes; Chronic diarrhea; severe associated disease;Taking antibiotics or probiotics in the last 3 months; Chronic inflammatory bowel disease; Weight ≤70Kg and hemoglobin level ≤7g/dl; Allergy to or refusal of any of the elements of the meal provided.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
Postprandial changes of plasma lipid fractions measured by lipidomic analysis and expressed as nmolof lipid/ml | Plasma samples will be collected at 2hours, 4hours, 6hours and 8hours after ingestion of the "western diet" meal to assess postprandial lipid fraction changes
  Lipidomic analysis of plasma lipid fractions expressed in ηm/ml after 12 hours of fasting and in the postprandial period (2h, 4h, 6h, 8h).

SECONDARY OUTCOMES:
Circulating markers of liver injury (AST, ALT, cytokeratin 18 fragments, microRNA-122) and serum cytokines (TNF-α, IL-6, IL-1β, IL-8). | After a 12hours overnight fast and then at 2, 4, 6 and 8hours after ingestion of the "western diet" meal.
  Circulating markers of liver injury (AST, ALT, cytokeratin 18 fragments, microRNA-122) and serum cytokines (TNF-α, IL-6, IL-1β, IL-8) will be measured after 12 hours of fasting and in the postprandial period (2h, 4h, 6h, 8h) in patients with NAFLD
Cytotoxic effect of postprandial plasma on hepatocytes in-vitro | Plasma samples at 2hours, 4hours, 6hours and 8hours after ingestion of the "western diet" meal.
  Hepatocytes will be cultured with postprandial plasma from NAFL or NASH patients, and incubated overnight. In-vitro hepatotoxicity will be evaluated using TUNEL assay, MTT assay and LDH release assay.
The effect of supernatants from hepatocyte cultures exposed to patient plasma on human macrophages in vitro | Plasma samples at 2hours, 4hours, 6hours and 8hours after ingestion of the "western diet" meal.
  Human macrophage will be cultured in vitro with supernatants from hepatocyte cultures exposed to patient plasma
Bacterial microbiome profiles | The day before or the morning before ingestion of the "western diet" meal.
  Bacterial microbiome profiles will be measured by the pyrosequencing technique of 16S RNA

CONTACTS AND LOCATIONS:
Overall Officials: Cosmin VOICAN, Principal Investigator — AP-HP, Beclere Hospital
Locations (1):
- Kremlin Bicetre hospital, Le Kremlin-Bicêtre, France